CLINICAL TRIAL: NCT04315194
Title: Efficacy of Clarithromycin-Naproxen-Oseltamivir Combination Therapy vs. Oseltamivir Alone for Hospitalised Paediatric Influenza Patients
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MackayMH
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Efficacy of Clarithromycin-Naproxen-Oseltamivir Combination Therapy vs. Oseltamivir Alone for Hospitalised Paediatric Influenza Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- clarithromycin-naproxen-oseltamivir: Efficacy of clarithromycin-naproxen-oseltamivir combination therapy vs. oseltamivir alone for hospitalised paediatric influenza patients
  Interventions: Drug: clarithromycin-naproxen-oseltamivir

INTERVENTIONS:
Drug: clarithromycin-naproxen-oseltamivir — to compare the safety and efficacy of clarithromycin-naproxen-oseltamivir combination therapy to that of oseltamivir treatment alone for hospitalised paediatric influenza patients.

SUMMARY:
Efficacy of clarithromycin-naproxen-oseltamivir combination therapy vs. oseltamivir alone for hospitalised paediatric influenza patients

DETAILED DESCRIPTION:
This study aimed to compare the safety and efficacy of clarithromycin-naproxen-oseltamivir combination therapy to that of oseltamivir treatment alone for hospitalised paediatric influenza patients. This prospective, single-blinded study included patients hospitalised for influenza infection aged 1 year to 18 years, at MacKay Children's Hospital, Taiwan, between December 2017 and December 2019. The primary outcomes were respiratory symptom severity and the signs that presented within hospitalisation. The durations of fever and hospital stay were also documented. The secondary outcome measures were serial changes in the virus titres, as detected by real-time polymerase chain reaction. Totally 54 patients were enrolled (28 in the control group and 26 in the combination group). There were no differences in the patients' baseline characteristics between the groups. The time to defervescence was significantly shorter in the combination group than the oseltamivir group (13.2 hours vs 32.1 hours, p=0.002). The decrease in the virus titre was more pronounced from days 1 to 3 (log Δ13) in the combination group than the oseltamivir group.(log Δ13: 39% vs 19%, p=0.001). In paediatric settings, combination therapy may be used selectively among patients with a history of febrile convulsion or families anxious about the discomforts associated with the fever itself.

ELIGIBILITY:
Inclusion Criteria:

- age 1 year to 18 years; body temperature higher than 38 °C; presence of one of the following symptoms-cough, sputum production, sore throat, rhinorrhoea, myalgia, headache, or fatigue presenting within 72 hours from symptom onset; laboratory-confirmed influenza infection (including rapid test or PCR-confirmed influenza A or B); and clinical requirement for hospitalisation. Antiviral treatment was initiated within 48 hours after admission.

Exclusion Criteria:

- a history of allergy or contraindication to the study medications; the administration of medications with macrolides (ex: azithromycin, erythromycin), naproxen or neuraminidase inhibitor use within 72 hours; current use of any antibiotic; and the presence of an immunocompromised state due to steroid use, human immunodeficiency virus infection, chronic kidney disease, renal failure, chemotherapy or radiotherapy in half year, or innate immunodeficiency.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study was conducted at Mackay Children's Hospital, Taiwan, between December 2017 and December 2019.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
severity of symptoms and signs | 1 month
  severity of symptoms and signs presenting on the first, third, and fifth days of admission, including cough, sputum, rhinorrhoea, sore throat, chills, wheezing/stridor, headache, dizziness, shortness of breath, chest pain, vomiting, diarrhoea, muscle pain, and abdominal pain. The duration of fever and length of hospital stay after treatment were also documented.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Wei Lee, Dr., Principal Investigator — Mackay Children's Hospital
Locations (1):
- Mackay Children's Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The data used to support the findings of this study have not been made available due to legal restrictions imposed by the government of Taiwan in relation to the "Personal Information Protection Act", personal data cannot be made publicly available. However, the investigators could provide disconnected data as follows:
  https://drive.google.com/open?id=1zcCZKNBO7kfJFt8AcuZd1Yi2PniAAlwe